CLINICAL TRIAL: NCT05660876
Title: Fistulotomy Versus Fistulotomy With Marsupialization, a Randomized Controlled Trial
Brief Title: Fistulotomy Versus Fistulotomy With Marsupialization
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: DHQ mardan (Other)
Responsible Party: Principal Investigator, Sajid Ali,FCPS, Consultant General surgeon, DHQ mardan
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 188-40
Record Dates: First submitted 2022-12-06; First posted 2022-12-21 (Actual); Last update posted 2022-12-21 (Actual); Status verified 2022-12

CONDITIONS: Fistula in Ano
MeSH Terms: conditions — Rectal Fistula

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Fistulotomy (Other): Standard fistulotomy was done in this arm
  Interventions: Procedure: standard fistulotomy; Procedure: fistulotomy with marsupialization
- Fistulotomy with marsupialization (Other): This arm consists of fistulotomy in which marsupialization was done
  Interventions: Procedure: standard fistulotomy; Procedure: fistulotomy with marsupialization

INTERVENTIONS:
Procedure: standard fistulotomy — in a standard manner fistula tract was identified and laid open without doing marsupialization
Procedure: fistulotomy with marsupialization — in this arm fistulotomy was done in a standard manner and marsupialization was done

SUMMARY:
It was a study comparing two standard procedures for fistula in ano

DETAILED DESCRIPTION:
It was a study which compared two standard surgical procedures for fistula in ano

ELIGIBILITY:
Inclusion Criteria:

* having low lying anal fistula Willing to enroll in study

Exclusion Criteria:

* unfit pts Having uncontrolled diabetes

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 60 (Actual)
Dates: Start 2020-08-01 (Actual); Primary Completion 2021-09-30 (Actual); Study Completion 2021-09-30 (Actual)

PRIMARY OUTCOMES:
Comparison of healing time in fistula in ano with and without marsupialization | 1year
  We measured the healing time between two groups

CONTACTS AND LOCATIONS:
Locations (1):
- Dhq, Mardan, Kpk, Pakistan

IPD SHARING:
Plan to Share IPD: No